CLINICAL TRIAL: NCT00898690
Title: Determination Of FEZ1/LZTS1 Expression As A Predictor Of Response To Taxol
Brief Title: Gene Expression in Predicting Response to Paclitaxel in Patients With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000355163; TJUH-02U.536
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2006-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cytogenetic Analysis; Gene Expression Profiling; Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction; Immunohistochemistry

INTERVENTIONS:
Genetic: cytogenetic analysis
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: mutation analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: immunohistochemistry staining method

SUMMARY:
RATIONALE: DNA analysis of tumor tissue may help doctors predict how patients who receive paclitaxel will respond to treatment.

PURPOSE: This laboratory study is evaluating gene expression in predicting response to paclitaxel in patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether loss of function of the FEZ1/LZTS1 gene is a predictor of response in patients with breast cancer treated with paclitaxel.

OUTLINE: This is a single-blind study.

Tumor tissue is analyzed for FEZ1/LZTS1 gene expression by immunohistochemistry using an antibody for the gene. Tumor expression of the gene is characterized by immunohistochemistry and scored by intensity of staining, percent of cell staining, and staining index. Tumor tissue is also analyzed for FEZ1/LZTS1 gene disruption by reverse transcriptase-polymerase chain reaction and direct sequencing.

PROJECTED ACCRUAL: Approximately 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer
* Measurable disease

  * Metastatic disease identified by imaging studies OR a primary disease site that will be treated in a neoadjuvant protocol
  * Lesions ≥ 10 mm by spiral CT scan
* Tumor tissue from the primary or metastatic site available for analysis by immunohistochemistry
* Previously treated OR planning to undergo treatment with paclitaxel* NOTE: *Concurrent enrollment on ECOG-2100 allowed
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2003-03

PRIMARY OUTCOMES:
Evaluation of the association between tumor expression of FEZ1/LZTS1 gene and response to paclitaxel

SECONDARY OUTCOMES:
Utility of FEZ1/LZTS1 gene expression in predicting the full 4-level response pattern (complete response, partial response, stable disease, progressive disease)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo M. Croce, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University